CLINICAL TRIAL: NCT03620396
Title: Comparison of Serum Levels of Trefoil Factor 3 in Patients With Gingivitis and Periodontitis Following Non Surgical Periodontal Therapy
Brief Title: Comparison of Serum Trefoil Factor 3 in Patients With Gingivitis and Periodontitis After Scaling and Root Planing
Acronym: CSTF3PGPSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.K.Sai Priyanka (Other)
Collaborators: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Sponsor-Investigator, Dr.K.Sai Priyanka, Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Organization: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Panineeya Mahavidyalaya; D159206045 (Other: Dr.NTR University of Health Sciences)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Gingivitis and Periodontal Diseases
MeSH Terms: conditions — Gingivitis; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: Patients will be equally divided into two test groups.Group A consists of Gingivitis patients and Group B consists of Periodontitis patients. Both the group patients have been evaluated for Serum Trefoil factor 3 at baseline and treated with non surgical periodontal therapy. After three months both the group patients were again assessed for serum trefoil factor 3.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Interventional (Experimental): Group A patients consists of Gingivitis patients whose serum is collected at base line and treated with Scaling and root planing and after three months serum is collected for assessment of Trefoil factor 3.
  Interventions: Procedure: Scaling and root planing
- Experimental Interventional (Experimental): Group B patients consists of Periodontitis patients whose serum is collected at base line and treated with Scaling and Root Planing and after three months serum is collected for assessment of Trefoil factor 3.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — After the serum collection is done from the patient for the assessment of trefoil factor 3, Non surgical periodontal therapy is carried out.

SUMMARY:
This study is intended to measure serum trefoil factor 3 at baseline and 3 months after, following nonsurgical periodontal therapy in patients with Gingivitis and Chronic Periodontitis.

DETAILED DESCRIPTION:
A goal of periodontal diagnostic procedure is to provide useful information to the clinician regarding the present periodontal disease type and severity. Advances in diagnostic research are moving towards methods where periodontal risk can be identified and quantified by objective measures such as Biomarkers.

Trefoil factors (TFFs) are one such secreted molecules derived from mucin producing epithelial cells of the gastro intestinal tracts and other tissues such as Salivary glands, Parotid ducts and oral mucosa. Among three Trefoil factors reported, Trefoil Factor 3 (TFF3) is the modifying factor for signalling pathway involved in cell survival, cell proliferation and cell migration of oral keratinocytes. Hence assessing the marker levels would achieve beneficial effects on diagnosing the disease severity.

ELIGIBILITY:
Inclusion Criteria:

For Gingivitis:

* Gingival Index: 1.1 to 2.
* Modifies Plaque Index: 1.0 to 1.9

For Periodontitis:

* Gingival Index: 1.1 to 2.
* Modifies Plaque Index: 1.0 to 1.9
* Probing depth > 4mm
* Clinical attachment loss > 2mm

Exclusion Criteria:

For Gingivitis:

* Presence of gingival recession.
* Presence of clinical attachment loss.
* Presence of furcation.
* Presence of systemic infections like diabetes, infections.
* Smokers.
* Antibiotic therapy received preceding 3 months.
* Patients who underwent periodontal therapy within 3 months.
* Pregnant and Lactating women.

For Periodontitis:

* Presence of any systemic conditions like diabetes, infections.
* Smokers.
* Antibiotic therapy received preceding 3 months.
* Patients who underwent periodontal therapy within 3 months.
* Pregnant and Lactating women.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-02-19 (Actual)

PRIMARY OUTCOMES:
Trefoil factor 3 | 3 months.
  Blood samples were collected by venepuncture of anti-cubital vein. 2ml of blood was collected in each test tube. 10 minutes after collection, the test tube containing 2ml blood was subjected to centrifugation at 3000rpm for 10 min. The supernatant straw colored fluid (serum) was separated into storage vials (Eppendorf tubes) for serum Trefoil Factor 3.

SECONDARY OUTCOMES:
Change in the Gingival Index. | 3 months
  The severity of gingivitis is scored on all surfaces of selected teeth using Williams Periodontal probe.
  Index teeth- 16, 12, 24, 36, 32, 44. Score around each tooth is totalled and divided by 4-score of tooth. 0.1-1.0: Mild gingivitis. 1.1-2.0:Moderate gingivitis 2.1-3.0:Severe gingivitis
Change in Modified Plaque Index | 3 months
  Examination of all the surfaces of the teeth are done using an explorer. The scores for individual teeth may be grouped and totalled and divided by the number of teeth.
  Excellent:0 Good:0.1-0.9 Fair:1.0-1.9 Poor:2-3
Change in Probing depth | 3 months
  The distance from the gingival margin to the depth of the pocket is measured using Williams periodontal probe.
Change in Clinical Attachment loss | 3 months
  The distance from the cementoenamel junction to the tip of the alveolar crest is measures using Williams periodontal probe.

REFERENCES:
- [Background] Chaiyarit P, Chayasadom A, Wara-Aswapati N, Hormdee D, Sittisomwong S, Nakaresisoon S, Samson MH, Pitiphat W, Giraud AS. Trefoil factors in saliva and gingival tissues of patients with chronic periodontitis. J Periodontol. 2012 Sep;83(9):1129-38. doi: 10.1902/jop.2011.110431. Epub 2011 Dec 19. PMID 22181686
- [Background] Storesund T, Schreurs O, Messelt EB, Kolltveit KM, Schenck K. Trefoil factor family 3 expression in the oral cavity. Eur J Oral Sci. 2009 Dec;117(6):636-43. doi: 10.1111/j.1600-0722.2009.00679.x. PMID 20121925